CLINICAL TRIAL: NCT05893849
Title: A Single Center, Open Label Study of Pharmacokinetics of Clinical Probes and Characteristics of Endogenous Biomarker for Drug-metabolizing Enzymes and Transporters in Chinese Older Adults
Brief Title: Pharmacokinetics of Clinical Probes and Characteristics of Endogenous Biomarker in Chinese Older Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dongyang Liu, Deputy Director Drug Clinical Trial Center, Peking University Third Hospital
Other Study IDs: M2022778
Record Dates: First submitted 2023-03-16; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Aging
Keywords: Chinese older adults; clinical probes; endogenous biomarkers; drug metabolizing enzymes; drug transporters

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older adults: Aged 60-74 years old, takes omeprazole or rabeprazole or pantoprazole or metoprolol or carvedilol or amlodipine or finasteride or simvastatin or rivaroxaban or meropenem or atorvastatin or rosuvastatin or metformin
  Interventions: Drug: Clinical probes
- Old older adults: Aged >75 years old, takes omeprazole or rabeprazole or pantoprazole or metoprolol or carvedilol or amlodipine or finasteride or simvastatin or rivaroxaban or meropenem or atorvastatin or rosuvastatin or metformin
  Interventions: Drug: Clinical probes

INTERVENTIONS:
Drug: Clinical probes — Inpatients taking one or more clinical probes of CYP2C19 (omeprazole, rabeprazole, pantoprazole), CYP2D6 (metoprolol, carvedilol), CYP3A4 (rivaroxaban, finasteride, amlodipine, simvastatin), OAT (meropenem), OATP1B1 (atorvastatin, rosuvastatin) and OCT (metformin) will be included in the study.

SUMMARY:
The goal of this observational study aims to reveal the pharmacokinetics of clinical probes and characteristics of endogenous biomarkers for drug-metabolizing enzymes and transporters in Chinese older adults and old older adults, to analyze their correlation with frailty, and to explore the exosome characteristics in this population.

DETAILED DESCRIPTION:
This study is a non-intervention observational study in Chinese older adults and will not interfere with the routine medical treatment. 6-10 mL whole blood and 20 mL urine samples (only applicable for patients taking meropenem and metformin) will be collected from eligible subjects according to medical routine blood collection time. Concentration of clinical probes and respective metabolites (when required), endogenous biomarkers, genotype information of drug-metabolizing enzymes and transporters, and the exosome characteristics will be quantified or measured.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults males and females aged 60-74 years old (older adults group) and ≥75 years old (old older adults group), proportion of either sex must not be less than 1/3 (except for subjects taking finasteride), number of subjects in each frailty category must not be less than 10;
2. Male participants must weight ≥45 kg and female participants must weight ≥40 kg. Body mass index (BMI) must be within the range of 18.0-28.0 (inclusive). BMI = weight (kg)/height^2 (m^2);
3. Inpatients with stable underlying disease, who takes any one or more of the following clinical probes: omeprazole/rabeprazole/pantoprazole/metoprolol/carvedilol/rivaroxaban/amlodipine/finasteride/simvastatin/meropenem/atorvastatin/rosuvastatin/metformin;
4. Creatinine clearance (CRCL) ≥15 mL/min, calculated by CockCroft-Gault equation. CRCL = [(140-age)*(lean body weight, kg)*(0.85 if female)/(72*Scr, mg/dL);
5. Willingness to comply with the study protocol and sign informed consent form.

Exclusion Criteria:

1. Subjects with known history of blood phobia or needle phobia that would preclude safe participation in the study procedures.
2. History of disease or an emerging disease within the past 1 month that could affect the study: Diseases affecting the abundance and activity of liver drug enzymes or transporters: cancer, diabetes (except metformin group), acute kidney injury, liver disease (cirrhosis, liver cancer, severe liver injury, severe fatty liver, liver abscess, internal bile duct stones, etc.)
3. History of major diseases or newly discovered diseases: prostate cancer, leukemia, liver cancer, breast cancer, colorectal cancer, leukemia and other tumor diseases;
4. Drugs that may affect the study were consumed within 1 week prior to screening:

   * Patients taking omeprazole/rabeprazole/pantoprazole: Potent CYP2C19 inhibitors: ASP8477, fluconazole, fluoxetine, fluvoxamine, ticlopidine; Potent CYP2C19 inducers: apalutamide, rifampicin, ritonavir;
   * Patients taking metoprolol/carvedilol: Potent CYP2D6 inhibitors: ASP8477, bupropion, fluoxetine, paroxetine, quinidine
   * Patients taking rivaroxaban/amlodipine/finasteride/simvastatin/atorvastatin: Potent CYP3A inhibitor: boceprevir, ceritinib, conivaptan hydrochloride, verapamil, diltiazem, aprepitant, quinidine, dronedarone, tacrolimus, protease inhibitors (ritonavir, indinavir, nelfinavir, saquinavir, lopinavir), macrolides antibiotics (erythromycin, clarithromycin, telithromycin), chloramphenicol, antifungal drugs (ketoconazole, itraconazole, posaconazole, voriconazole, fluconazole, miconazole) nefazoldone, cobistat, cimetidine, ciprofloxacin, fluvoxamine, imatinib, St. John's wort, ranolazine; Potent CYP3A inducers: apalutamide, avomibe, rifampicin, carbamazepine, enzalutamide, ivosidenib, mitotane, phenytoin, rifapentine
   * Patients taking meropenem: Potent OAT inhibitors: aminohippuric acid, probenecid, teriflunomide
   * Patients taking simvastatin/atorvastatin/rosuvastatin: Potent OATP1B1 inhibitor: protease inhibitor (atazanavir, ritonavir, lopinavir, simeprevir), cyclosporin, macrolides antibiotics (erythromycin, clarithromycin), rifampicin;
5. Subjects who have smoking addict or alcohol abuse and do not agree to abstain from smoking or drinking during the trial period (smoking addict: average of ≥5 cigarettes daily; alcohol abuse: average of ≥100mL hard liquor);
6. Tested positive on virological test (human immunodeficiency virus antibody (HIV-Ab)), syphilis serological test, hepatitis B virus surface antigen (HBsAg), or hepatitis C virus antibody (HCV-Ab) within 6 months prior to screening;
7. Subjects who have participated in clinical trials of any drug or medical device within 3 months prior to screening;
8. Subjects who have any factors deemed unsuitable for participation in this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients aged 60-74 years old (older adults group) and ≥75 years old (old older adults group) with stable underlying disease, takes any one or more of the following clinical probes: omeprazole/rabeprazole/pantoprazole/metoprolol/carvedilol/rivaroxaban/amlodipine/finasteride/simvastatin/meropenem/atorvastatin/rosuvastatin/metformin.
Sampling Method: Non-Probability Sample
Enrollment: 624 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Concentration of clinical probes in plasma | Sampling will be performed according to routine medical follow-up, which should be no less than 3 samples over the period of one year
  Plasma concentration of clinical probes and the respective metabolites (when required) will be quantified and measured by LC-MS/MS or HPLC
Concentration of clinical probes in urine | Urine samples will be collected at any administration intervals, which should be no less than 1 sample over the period of one year
  Urine concentration of meropenem and metformin will be quantified and measured by LC-MS/MS or HPLC
Level of endogenous biomarker | sampling will be performed according to routine medical follow-up, which should be no less than 3 samples over the period of one year
  The level of endogenous biomarker (Dihydroxyeicosatrienoic acids, DHETs, 4β-hydroxycholesterol/cholesterol ratio, 4β-OHC/CHO, pyridoxic acids, PDA, Coproporphyrin, CP) will be quantified and measured by LC-MS/MS or HPLC or ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang Liu, Principal Investigator — Drug Clinical Trial Center
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No